CLINICAL TRIAL: NCT04079387
Title: Effect of Endotracheal Tube Plus STYLET Versus Endotracheal Tube Alone on Successful First-Pass Orotracheal Intubation Among Critically Ill Patients: the Randomised STYLETO Study Protocol"
Brief Title: Effect of Endotracheal Tube Plus STYLET Versus Endotracheal Tube Alone
Acronym: STYLETO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0216
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Intubation Complication; Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENDOTRACHEAL TUBE + STYLET (Experimental): The experimental group consists in intubating the trachea with an endotracheal tube + stylet with a "straight-to-cuff" shape and a bend angle of 25° to 35°.
  Interventions: Device: ENDOTRACHEAL TUBE + STYLET
- ENDOTRACHEAL TUBE ALONE (Active Comparator): The control group consists in intubating the trachea with an endotracheal tube alone (i.e, without stylet).
  Interventions: Device: ENDOTRACHEAL TUBE ALONE

INTERVENTIONS:
Device: ENDOTRACHEAL TUBE + STYLET — The experimental group consists in intubating the trachea with an endotracheal tube + stylet with a "straight-to-cuff" shape and a bend angle of 25° to 35°
  Arms: ENDOTRACHEAL TUBE + STYLET
Device: ENDOTRACHEAL TUBE ALONE — intubating the trachea with an endotracheal tube alone
  Arms: ENDOTRACHEAL TUBE ALONE

SUMMARY:
Patients admitted to Intensive Care Units (ICU) often require respiratory support. Orotracheal intubation is one of the most frequent procedures performed in ICU.When performed in emergency settings, intubation is a challenging issue as it may be associated with life-threatening complications in up to one third of cases

Using a preshaped endotracheal tube plus stylet may have potential advantages over endotracheal tube alone without stylet. The stylet is a rigid but malleable introducer which fits inside the endotracheal tube and allows for manipulation of the tube shape; usually into a hockey stick shape, to facilitate passage of the tube through the laryngeal inlet. The stylet can help to increase success of intubation in operating rooms

DETAILED DESCRIPTION:
Patients admitted to Intensive Care Units (ICU) often require respiratory support. Orotracheal intubation is one of the most frequent procedures performed in ICU. When performed in emergency settings, intubation is a challenging issue as it may be associated with life-threatening complications in up to one third of cases.Severe hypoxaemia occurring during intubation procedure can result in cardiac arrest,cerebral anoxia, and death.Difficult intubation is known to be associated with life-threatening complications both in operating room and in emergent conditions.ICU intubation conditions are worse than intubation conditions in operative rooms.A non-planned and urgent intubation procedure, severity of patient disease and ergonomic issues explain the morbidity associated with intubation in ICU.To prevent and limit the incidence of severe hypoxemia following intubation and its complications, several intubation algorithms have been developed ,and specific risk factors for difficult intubation in ICU have been identified.

In 2018, a large multicenter study reported first-attempt intubation success rates using direct laryngoscopy of 70% and videolaryngoscopy of 67%. In 2019, a multicentre randomized trial,assessing whether positive-pressure ventilation with a bag-mask device (bag-mask ventilation) during tracheal intubation of critically ill adults prevents hypoxemia, reported a first-attempt success rate of 81%. Other authors reported an overall first-attempt intubation success rate of 74%. The 20% to 40% first-attempt failure rates throughout studies highlight the opportunity to improve the safety and efficiency of this critical procedure. Using a preshaped endotracheal tube plus stylet may have potential advantages over endotracheal tube alone without stylet. The stylet is a rigid but malleable introducer which fits inside the endotracheal tube and allows for manipulation of the tube shape; usually into a hockey stick shape, to facilitate passage of the tube through the laryngeal inlet. The stylet can help to increase success of intubation in operating rooms.

However, some complications from intubating stylets have been reported including mucosal bleeding, perforation of the trachea or esophagus, and sore throat. In 2018, one study has assessed the effect of adding a stylet in case of difficult intubation in prehospital setting.However, in ICU, the systematic use of a stylet is still debated and recent recommendations do not recommend to use or not to use such devices for first-pass intubation. The device chosen for intubation may therefore be a confounding factor between the relation of stylet use and first-attempt success.The routine use of a stylet for first-pass intubation using laryngoscopes in ICU has never been assessed and benefit remains to be established.

The investigators hypothesis that adding stylet to endotracheal tube will increase the frequency of successful first-pass intubation compared with use endotracheal tube alone (i.e, without stylet) in ICU patients needing mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be present in the intensive care unit (ICU) and require mechanical ventilation through an orotracheal tube.
* Adult (age ≥ 18 years)
* Subjects must be covered by public health insurance
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Refusal of study participation or to pursue the study by the patient
* Pregnancy or breastfeeding
* Absence of coverage by the French statutory healthcare insurance system
* protected person
* intubation in case of cardio circulatory arrest
* Previous intubation during the same ICU stay and already included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with successful first-pass orotracheal intubation | At intubation
  the proportion of patients with successful first-pass orotracheal intubation

SECONDARY OUTCOMES:
Complications related to intubation | 1 hour after intubation
  severe hypoxemia defined by lowest oxygen saturation (SpO2) < 80 %, severe cardiovascular collapse, defined as systolic blood pressure less than 65 mm Hg recorded at least once or less than 90 mm Hg lasting 30 minutes despite 500-1,000 ml of fluid loading (crystalloids solutions) or requiring introduction or increasing doses by more than 30% of vasoactive support, cardiac arrest, death during intubation; moderate: difficult intubation, severe ventricular or supraventricular arrhythmia requiring intervention, oesophageal intubation, agitation, pulmonary aspiration, dental injuries

OTHER OUTCOMES:
Lowest SpO2 up to 24 hours after intubation | up to 24 hours after intubation
  Assessment of the value of the lowest SpO2
Highest positive end expiratory pressure (PEEP) up to 24 hours after intubation | up to 24 hours after intubation
  Assessment of the value of the highest PEEP
Highest fraction of inspired oxygen (FiO2) up to 24 hours after intubation | up to 24 hours after intubation
  Assessment of the value of the highest FiO2
lowest SpO2 < 90% | during intubation
  incidence of lowest SpO2 less than 90% from induction to 2 minutes after intubation
Change in SpO2 | during intubation
  Change in SpO2 from SpO2 at induction to lowest SpO2
desaturation | during intubation
  desaturation, defined as a change in SpO2 of more than 3% from induction to 2 minutes after intubation
Cormack Lehane | during intubation
  Cormack-Lehane grade of glottic view
difficulty of intubation | during intubation
  operator-assessed difficulty of intubation
additional airway equipment or second operator | during intubation
  need for additional airway equipment or a second operator
laryngoscopy attempts | during intubation
  number of laryngoscopy attempts
Lowest SpO2 from 0-1 hour post intubation | up to 1 hour after intubation
  Assessment of the value of the lowest SpO2 from 0-1 hours after intubation
Highest FiO2 from 0-1 hour post intubation | up to 1 hour after intubation
  Assessment of the value of the highest FiO2 from 0-1 hours after intubation
Highest PEEP from 0-1 hour post intubation | up to 1 hour after intubation
  Assessment of the value of the highest PEEP from 0-1 hours after intubation
Lowest SpO2 from 1-6 hours post intubation | From 1 to 6 hours after intubation
  Assessment of the value of the lowest SpO2 from 1-6 hours after intubation
Highest FiO2 from 1-6 hours post intubation | From 1 to 6 hours after intubation
  Assessment of the value of the highest FiO2 from 1-6 hours after intubation
Highest PEEP from 1-6 hours post intubation | From 1 to 6 hours after intubation
  Assessment of the value of the highest PEEP from 1-6 hours after intubation
new infiltrate | Up to 48 hours after intubation
  new infiltrate on chest imaging in the 48 hours after intubation
new pneumothorax | Up to 24 hours after intubation
  new pneumothorax on chest imaging in the 24 hours after intubation
new pneumomediastinum | Up to 24 hours after intubation
  new pneumomediastinum on chest imaging in the 24 hours after intubation
Intensive care unit (ICU) length of stay | Up to 90 days after intubation
  ICU length of stay
ICU-free days | Up to 90 days after intubation
  ICU-free days
invasive ventilator-free days | Up to 90 days after intubation
  invasive ventilator-free days
mortality rate on day 28 | Up to 28 days after intubation
  mortality rate on day 28
In hospital mortality | Up to 90 days after intubation
  in hospital mortality
mortality rate on day 90 | Up to 90 days after intubation
  mortality rate on day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Montpellier, Saint Eloi, Montpellier, Languedoc-Roussillon, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and institutional review board (IRB) review. Dataset will be shared after careful examination by the study board of investigators.

REFERENCES:
- [Background] Jaber S, Rolle A, Godet T, Terzi N, Riu B, Asfar P, Bourenne J, Ramin S, Lemiale V, Quenot JP, Guitton C, Prudhomme E, Quemeneur C, Blondonnet R, Biais M, Muller L, Ouattara A, Ferrandiere M, Saint-Leger P, Rimmele T, Pottecher J, Chanques G, Belafia F, Chauveton C, Huguet H, Asehnoune K, Futier E, Azoulay E, Molinari N, De Jong A; STYLETO trial group. Effect of the use of an endotracheal tube and stylet versus an endotracheal tube alone on first-attempt intubation success: a multicentre, randomised clinical trial in 999 patients. Intensive Care Med. 2021 Jun;47(6):653-664. doi: 10.1007/s00134-021-06417-y. Epub 2021 May 25. PMID 34032882
- [Derived] Jaber S, Rolle A, Jung B, Chanques G, Bertet H, Galeazzi D, Chauveton C, Molinari N, De Jong A. Effect of endotracheal tube plus stylet versus endotracheal tube alone on successful first-attempt tracheal intubation among critically ill patients: the multicentre randomised STYLETO study protocol. BMJ Open. 2020 Oct 7;10(10):e036718. doi: 10.1136/bmjopen-2019-036718. PMID 33033014